CLINICAL TRIAL: NCT02017236
Title: A Single Center, Open-label, Randomized, Four-Sequence, Four-period Crossover Study to Investigate Food Effect on the Pharmacokinetics of Single Dose of Volitinib in Healthy Subjects
Brief Title: A Food Effect Phase I Study of the Volitinib in Healthy Subjects
Acronym: HMPL-504
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-504-CH1
Record Dates: First submitted 2013-11-27; First posted 2013-12-20 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2013-12

CONDITIONS: Food Effect; Health Subjects
Keywords: Food Effect; Health subjects
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volitinib ,after high fat meal intake (Experimental): A:single oral Volitinib after high fat meal intake
  Interventions: Drug: Volitinib
- Volitinib,after general diet (Experimental): B:single oral Volitinib, after general diet
  Interventions: Drug: Volitinib

INTERVENTIONS:
Drug: Volitinib — 600mg Volitinib ,single dose,oral
  Other Names: HMPL-504

SUMMARY:
The purpose of this study is to evaluate to determine the effect of food on the PK of a single dose of 600 mg Volitinib and its two major metabolites in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate to determine the effect of food on the PK( pharmacokinetics) of a single dose of 600 mg Volitinib and its two major metabolites in healthy subjects and to assess the safety and tolerability of single doses of 600mg in healthy subjects.This study will be an open-label, randomized, four-period, crossover PK food effect study of Volitinib administered orally at 600 mg. Subjects will be screened for eligibility up to 14 days prior to entry into the study,there will be 4 treatments,2 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males , between 18 and 45 years of age, inclusive.
* Body mass index (BMI) within the range of 19 to 25 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs.
* Adequate hepatic, renal, heart, and hematologic functions
* Male subjects who are either sterile or agree to use, during the period from informed consent until 90 days following Study Completion, 1 of the following approved methods of contraception: a double barrier method (eg, male condom with spermicide, use by female sexual partner of an intrauterine device with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, a diaphragm with spermicide, or use of a cervical cap with spermicide); a sterile sexual partner; a female sexual partner using an intravaginal system (eg,NuvaRing®); or a partner using an oral, implantable, transdermal, or injectable contraceptives.
* Able to comprehend and willing to sign an informed consent form (ICF).

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric disorder(as determined by the Investigator).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* History of stomach or intestinal surgery, nephrectomy, cholecystectomy or resection that would potentially alter absorption and/or excretion of orally administered drugs as determined by the investigator (appendectomy and/or hernia repair may be allowed).
* History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
* Diagnosis of alcoholism or drug addiction within 1 year prior to Period 1 Check-in.
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer prior to informed consent.
* Use of any prescription medications or products within 14 days prior to Period 1 prior to informed consent.
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic, herbal, dietary supplements, or plant derived preparations) within 7 days prior to each study period Check-in.
* Use of alcohol-, grapefruit-, Seville orange-, or caffeine-containing foods, juices, or beverages within 72 hours prior to each study period Check-in.
* Use of known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort, etc.) for a period of 60 days prior to informed consent;
* Poor peripheral venous access.
* Donation of blood ≥ 250 mL from 30 days prior to informed consent until study completion, inclusive, or of plasma from 2 weeks prior to informed consent until study completion, inclusive.
* Receipt of blood products within 2 months prior to Period 1 Check-in;
* Blood pressure greater than 140/90 mmHg confirmed by repeat at Screening or at Period 1 Check-in.
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 1-3days after every drug administration
  The following PK parameters will be derived from the plasma concentration-time profile of Volitinib following administration:Area Under Curve (AUC), both from time zero to time with last observation and from time zero to infinity;;Maximum plasma concentration (Cmax);Time to reach the Cmax (Tmax);Apparent oral Clearance (CL/F);Apparent oral Volume of distribution (Vz/F);Other parameters, such as elimination half-life

SECONDARY OUTCOMES:
Safety | 1 day to the 14days after every drug administration
  AE(adverse event) will be summarized by type and severity

OTHER OUTCOMES:
Urinal and fecal excretion ratio of Volitnib;renal clearance of Volitinib | duriation the first day to the third day after every drug administration
  Urinal and fecal excretion ratio of Volitnib, renal clearance of Volitinib;Preliminary metabolite profiling of Volitnib in healthy subjects, with preliminary understanding of the clearance mechanism of Volitinib in human

CONTACTS AND LOCATIONS:
Overall Officials: Chen yu, Principal Investigator — Xuhui Center Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China